CLINICAL TRIAL: NCT04997889
Title: Efficacy (Preliminary) and Safety of Artificial Salivary Containing Cumin and Ginger Extract in Healthy Volunteer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EC2105120
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Health, Subjective
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial salivary containing cumin and ginger extract (Experimental): The artificial salivary containing cumin and ginger extract will be used 2 g/time (3 times/day) into the mouth for 6 days. Then, the artificial salivary containing cumin and ginger extract will be stopped for 7-10 days. After that, the artificial salivary containing cumin and ginger extract will be used 2 g/time (3 times/day) into the mouth for 3 days.
  Interventions: Combination Product: Artificial salivary containing cumin and ginger extract
- Commercial artificial salivary (Active Comparator): The commercial artificial salivary will be used 2 g/time (3 times/day) into the mouth for 6 days. Then, the commercial artificial salivary will be stopped for 7-10 days. After that, the commercial artificial salivary will be used 2 g/time (3 times/day) into the mouth for 3 days.
  Interventions: Other: Commercial artificial salivary

INTERVENTIONS:
Combination Product: Artificial salivary containing cumin and ginger extract — The artificial salivary containing cumin and ginger extract will be used 2 g/time (3 times/day) into the mouth for 6 days. Then, the artificial salivary containing cumin and ginger extract will be stopped for 7-10 days. After that, the artificial salivary containing cumin and ginger extract will be used 2 g/time (3 times/day) into the mouth for 3 days.
  Arms: artificial salivary containing cumin and ginger extract
Other: Commercial artificial salivary — The commercial artificial salivary will be used 2 g/time (3 times/day) into the mouth for 6 days. Then, the commercial artificial salivary will be stopped for 7-10 days. After that, the commercial artificial salivary will be used 2 g/time (3 times/day) into the mouth for 3 days.
  Arms: Commercial artificial salivary

SUMMARY:
This study is a preliminary clinical study about safety of artificial salivary containing cumin and ginger extract in 21 healthy volunteers. After the preliminary clinical study, safety of artificial salivary containing cumin and ginger extract in 112 healthy volunteers. The volunteers will be divided into 2 groups which are artificial salivary containing cumin and ginger extract group and commercial artificial salivary.

DETAILED DESCRIPTION:
This study is a preliminary clinical study about safety of artificial salivary containing cumin and ginger extract in 21 healthy volunteers. The volunteers will be divided into 3 groups which are artificial salivary containing 0.3% cumin and 0.05%ginger extract group, artificial salivary containing 0.3%cumin and 0.1%ginger extract group, and artificial salivary containing 0.3%cumin and 0.15%ginger extract group. The volunteers will be evaluated salivary volume by Schirmer test, salivary acid and base value by strip test, dry mouth by questionnaire, and adverse effects before and after using the artificial salivary for 30 min. After the preliminary clinical study, safety of artificial salivary containing cumin and ginger extract in 112 healthy volunteers. The volunteers will be divided into 2 groups which are artificial salivary containing cumin and ginger extract group and commercial artificial salivary. The volunteers will be evaluated salivary acid and base value by strip test and adverse effects by World Health Organization Oral Mucositis Grading Scale and questionnaire before and after using the artificial salivary (3 times/day) for 3 and 6 days. Then, the volunteers will stop using the artificial salivary for 7-10 days. After that, the volunteers will be used the artificial salivary for 3 days. All evaluation will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* World Health Organization Oral Mucositis Grading Scale =0
* No using artificial salivary or activated salivary medicine more than 2 weeks
* No cumin, ginger, xylitol, glycerin allergy
* Have a willingness to participate in the study

Exclusion Criteria:

* Uncontrolled disease
* Dry mouth
* Salivary gland disease, inflammation, or sialolith
* Pregnancy or lactation
* During participated in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Salivary acid and base value | 6 days
  Salivary acid and base value (scale 0 (acid) to 14 (base)) using strip test

SECONDARY OUTCOMES:
Mucositis | 6 days
  Mucositis using World Health Organization Oral Mucositis Grading Scale (scale 0 (none) to 4 (life-threatening)
Adverse event | 6 days
  Adverse event using questionnaire (Yes or No)
Dry mouth status | 6 days
  Dry mouth status using questionnaire (scale 0 (none) to 10 (severe symptom)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand